CLINICAL TRIAL: NCT03446365
Title: Peer-Administered Asthma Self-Management Intervention in Urban Middle Schools
Acronym: PeerASMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R01MD012225-01 (NIH)
Record Dates: First submitted 2018-01-24; First posted 2018-02-26 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Asthma
Keywords: Asthma; Latino children; middle school; peer models; educational intervention; high school students
MeSH Terms: conditions — Asthma | interventions — Child Health

STUDY DESIGN:
Intervention Model Description: 6th to 8th grade middle schoolers will be enrolled then randomly assigned to one of three conditions: 1) ASMAS, 6th to 8th grade middle schoolers will be enrolled then randomly assigned to 1) ASMAS, or 2) Asthma Education plus Child Health control condition, or 3) a no treatment control condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASMAS (Experimental): ASMAS is an asthma self-management program based on NHLBI clinical guidelines for optimal school-based asthma management. It involves 4, 1½ hour sessions delivered in group format in the urban, middle school setting by a Latino High School Peer who has asthma. ASMAS focuses on asthma pathophysiology, symptom management, asthma medications, and trigger control.
  Interventions: Behavioral: ASMAS
- Asthma education plus child health (Active Comparator): Asthma Education plus Child Health control condition will be delivered by an adult Health Educator , and includes 4 sessions (1 1/2 hrs long) of our existing asthma education ("Asthma's Magic Number") with added general health topics (nutrition, physical activity, safety).
  Interventions: Behavioral: Asthma education plus child health
- No Treatment Control (No Intervention): Students randomly assigned to this arm , will receive standard of care, which is no treatment, and will not participate in any group intervention sessions.

INTERVENTIONS:
Behavioral: ASMAS — A high school peer led group intervention for middles school students targeting asthma education and asthma management practices.
  Arms: ASMAS
Behavioral: Asthma education plus child health — Health educator led intervention focused on asthma education and other child health topics.
  Arms: Asthma education plus child health

SUMMARY:
Health disparities in pediatric asthma persist, with Latino children demonstrating increased asthma morbidity. Middle school children with asthma have greater morbidity than children from any other age group and spend a majority of their day in school, where they must manage any asthma. The investigators developed and piloted a novel group-based intervention - ASMAS (Asthma Self-MAnagement in Schools) in two geographic areas with a high prevalence of urban and Latino children with asthma: Providence, Rhode Island, and San Juan, Puerto Rico. ASMAS is a 4-session, peer-facilitated asthma self-management intervention specific to the school setting for Latino middle school (6th-8th graders) children. It is delivered by trained High School Juniors and Seniors of Latino descent with asthma. The preliminary effects of ASMAS for improving asthma outcomes and self-management relative to controls were demonstrated in a previous intervention development study. This study will evaluate ASMAS through a large-scaled Randomized Control Trial with urban middle school students who have persistent asthma in Providence, Rhode Island and San Juan, Puerto Rico and will identify barriers and facilitators to the implementation of ASMAS. These results will inform future, large-scale dissemination in other urban school settings.

DETAILED DESCRIPTION:
The goal of this study is to evaluate a 4-session, peer-facilitated asthma self-management intervention for Latino, middle school (6th-8th) youth in urban public school settings. The intervention, ASMAS (Asthma Self-Management in Schools) is administered by trained and supervised High School juniors and seniors of Latino descent with asthma to middle school peers with asthma. This study is a partnership with a second research group in San Juan, Puerto Rico, since there is also a high rate of asthma in children there.

There are 2 goals in this study. The first goal is to evaluate the effects of ASMAS on asthma health outcomes (for example, asthma control, symptom free days, school absences and lung function) and on asthma self-management (skills, knowledge and self-efficacy, availability of rescue inhaler and action plan at school) in a sample of 432 Latino middle school children with asthma in Providence, Rhode Island and San Juan, Puerto Rico.

Middle schoolers and a primary caregiver will complete a baseline research session, as well as, immediately post intervention and 4-month, 8-month and 12-month post intervention follow-up research home visits during which they will complete study questionnaires about the child's asthma. Students will be randomly assigned to one of three study groups. Assignment is random (like a coin toss), and what each student does in school depends on what group each student is assigned to. The ASMAS group and the Asthma + Health Education groups will learn about asthma and about other selected health topics during their in-school intervention sessions (1 per week for 4 weeks). The "no treatment" study group will not attend in-school group sessions at all.

The second goal in the study is to evaluate the intervention in preparation for using it on a wider scale in other places. Students, caregivers, High School Peers, school administrators and additional community members will be invited to participate in group discussions about the intervention.

ELIGIBILITY:
Inclusion Criteria specify that students must:

* Be 11-14 years old
* Attend 6th, 7th or 8th grade
* attend a targeted public school
* have physician-diagnosed asthma according to caregiver and provider report
* meet criteria for current persistent asthma either by a) having a current prescription for an asthma controller medicine, or b) having any of the following in the previous 4 weeks:

I. daytime asthma symptoms > 2 days/week,

II. nighttime awakenings due to asthma at least 3-4 times/month,

III. short-acting beta agonist use at least 2 days/week,

IV. activity limitation, or

V. oral steroid use at least 2 times/year

* children must have recent active asthma activity in the previous 4 weeks through endorsement of any of criteria I-V above
* In Rhode Island, children's primary caregiver must identify as Latino
* In Rhode Island, children must speak English

Exclusion criteria:

* active immunotherapy,
* other pulmonary disease,
* receiving special education services in a self-contained classroom,
* any severe psychiatric or medical conditions

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 243 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in asthma control | Assessed at baseline, immediately post intervention, and 4 months post intervention , 8 months post intervention, and 12-months post intervention
  Assessed by child and parent report through the 7-item Child Asthma Control Test (C-ACT)
Change in symptom free days | Assessed at baseline, immediately post intervention, and 4 months post intervention , 8 months post intervention, and 12-months post intervention
  By parent report using standard questionnaire of symptom-free days/nights in prior 30 days
Change in asthma related school absence ratio | Assessed at baseline, immediately post intervention, and 4 months post intervention , 8 months post intervention, and 12-months post intervention
  Asthma related school absence ratio will be calculated from school attendance data and caregiver report of school absences due to asthma
Change in lung function | Assessed at baseline, immediately post intervention, and 4 months post intervention , 8 months post intervention, and 12-months post intervention
  The Asthma Monitor 2 (AM2, ERT, USA) is a hand-held, computerized spirometer that collects pulmonary function indexes (Forced Expiratory Volume at one second, FEV1 ). Children will use AM2 during one week using standard procedures, 2x/day (before medications AM/PM). FEV1 predicted will be obtained.

SECONDARY OUTCOMES:
Change in child asthma knowledge | Assessed at baseline, immediately post intervention, and 4 months post intervention , 8 months post intervention, and 12-months post intervention
  Child report through the valid and reliable Asthma Knowledge Questionnaire
Change in child asthma self-efficacy | Assessed at baseline, immediately post intervention, and 4 months post intervention , 8 months post intervention, and 12-months post intervention
  Child report through valid and reliable children's Asthma Self-Efficacy Scale (Cronbach alpha .87; Bursch, et al, 1999). The scale includes 14 items with responses ranging from 1 to 6, and higher scores indicate more self-efficacy to care for asthma. An asthma self-efficacy score is calculated using the average of the 14 items.
Change in asthma self-management | Assessed at baseline, immediately post intervention, and 4 months post intervention , 8 months post intervention, and 12-months post intervention
  Through a well-validated and reliable measure; child and caregiver versions
Change in asthma Action plan/Inhaler availability | Assessed at baseline, immediately post intervention, and 4 months post intervention , 8 months post intervention, and 12-months post intervention
  School Nurse report of Availability of rescue inhaler at school and asthma action plan with school nurse

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Koinis-Mitchell, PhD, Principal Investigator — Rhode Island Hospital; Glorisa Canino, PhD, Principal Investigator — University of Puerto Rico; Sheryl J Kopel, MSc, Study Director — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No